CLINICAL TRIAL: NCT01621555
Title: Pain Sensitivity and Outcome in Arthroscopic Shoulder Surgery
Acronym: PSOASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Fife (Other Government)
Responsible Party: Principal Investigator, Tony Davis, Dr Anthony Davis, NHS Fife
Other Study IDs: PSOASS1
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Anomaly; Shoulder
Keywords: shoulder surgery; Pain sensitivity; Rowe score; Constant Score; Surgical Outcome; Postoperative pain
MeSH Terms: conditions — Congenital Abnormalities; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PSOASS Patients: Patients undergoing elective arthroscopic shoulder surgery

SUMMARY:
The purpose of this study is to investigate whether there is a correlation between a patients pain sensitivity and their subsequent post-operative pain and surgical outcome in arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Arthroscopic shoulder surgery is increasingly performed on a daycase basis. Optimal pain relief is the goal as this not only improves patient comfort and allows expedient discharge from hospital, but also reduces the risk of developing postoperative chronic pain and may improve surgical outcome. However, optimal postoperative pain control in daycase surgery remains a challenge. There is considerable variation in the level of postoperative pain experienced between individuals and subsequent analgesia requirements. Previous studies have attempted to predict the level of postoperative pain an individual will experience, using a variety of complex preoperative pain and psychological assessments. Other investigators have focused on a simpler approach, by testing an individual's pain threshold to a single preoperative nociceptive (painful) stimulus, e.g. heat or pressure. Recent work has produced a simple questionnaire alternative to pain intensity testing, the Pain Sensitivity Questionnaire (PSQ). We hypothesise that a patient's pain sensitivity preoperatively may both affect the level of pain they experience postoperatively and their final surgical outcome.

The aim of our study is to correlate a patient's pain sensitivity, as measured by the Pain Sensitivity Questionnaire, with the degree of acute postoperative pain (first 4 days) they experience and subsequent surgical outcome at 6 months.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 years or older, attending for arthroscopic shoulder surgery (stabilisation, rotator cuff repair, arthrolysis, subacromial decompression), able to give informed consent.

Exclusion Criteria:

* Unable to give informed consent
* Documented sensory abnormality (e.g. peripheral neuropathy)
* Contraindication to proposed anaesthetic/analgesic regimen
* No telephone or unable to communicate in English
* Documented psychiatric disorder
* Documented/suspected substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting for elective arthroscopic shoulder surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Degree of correlation between Pain Sensitivity Questionnaire score and 6 month postoperative Rowe/Constant Score. | 6 months

SECONDARY OUTCOMES:
The degree of correlation between Pain Sensitivity Questionnaire scores and 'Area Under the Curve (AUC)' for postoperative pain experienced (generated from the VAS scores over 4 postoperative days). | 6 months
• The degree of correlation between AUC for postoperative pain and 6 month Constant/Rowe score. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ANTHONY H DAVIS, MBCHB FRCA, Principal Investigator — NHS Fife
Locations (1):
- NHS FIFE, Kirkcaldy, Fife, United Kingdom